CLINICAL TRIAL: NCT01521754
Title: Medtronic Registry for Epilepsy (MORE)
Brief Title: Product Surveillance Registry- Deep Brain Stimulation for Epilepsy
Acronym: MORE
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1.02.9001; Addendum C.AD.1 (Other: Addendum C.AD.1)
Record Dates: First submitted 2012-01-13; First posted 2012-01-31 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Perspective: Prospective cohort: new patients who are initially implanted with a Medtronic neurostimulation system on or after a site's activation date. The classification is static and will not change in the case of a re-implant.
- Retrospective: Retrospective cohort: existing patients comprised the sub-group of patients who were implanted with a Medtronic neurostimulation system prior to a site's activation date. This cohort contains a part of retrospective data and a part of prospective data according to the enrolment date. The classification is static and will not change even when an existing patient will be subsequently re-implanted after the site's activation date.

SUMMARY:
The purpose of this observational registry is to evaluate the long-term effectiveness, safety and performance of market-released Medtronic Neuromodulation products for Deep Brain Stimulation (DBS) for the treatment of refractory epilepsy. In addition, healthcare resource use and patient reported outcomes, such as health related quality of life will be assessed.

DETAILED DESCRIPTION:
Introduction

The purpose of this observational registry is to evaluate the long-term effectiveness, safety and performance of market-released Medtronic Neuromodulation products for Deep Brain Stimulation (DBS) for the treatment of refractory epilepsy. In addition, healthcare resource use and patient reported outcomes, such as health related quality of life will be assessed.

Enrollment and Duration Patients meeting the eligibility criteria for the implantation of the Medtronic® DBS™ Therapy for Epilepsy will be included in the registry. Approximately 200 patients meeting all the eligibility criteria will be prospectively enrolled over an expected two-year period.

Approximately 30 centers, mainly from across Europe will participate. Center selection could also be extended to sites outside Europe.

Each patient will perform follow-up visits according to clinical practice.

The estimated duration of the registry will be approximately 49 months (24 months for the enrollment phase, 24 months for follow-up visits and 1 month for final data collection).

Inclusion and exclusion criteria Inclusion criteria

* Fulfilling the criteria of labeling indications of Medtronic® DBS™ Therapy for Epilepsy.
* Patient with diagnosis of refractory epilepsy as defined by 1981 ILAE (International League Against Epilepsy) classification, who have been implanted or will be implanted with Medtronic® DBS™ Therapy for Epilepsy.
* For both cohorts, completed at least two full consecutive months diary information on seizure type and frequency prior to DBS implant (seizure type should be classified at least as simple partial, complex partial, partial evolving to secondarily generalized seizures, and generalized). In regard to the prospective cohort, the patient will be conditionally enrolled at the enrolment visit, and the criterion will be reassessed at the baseline visit.
* Patient or patient's legally authorized representative able to understand and to provide written informed consent and/or authorization for access to and use of health information, as required by an institution's IRB/MEC or local law and regulations.

Exclusion criteria

* Incomplete and/or unreliable patient seizure diary based on the physician's judgment
* Patient is currently enrolled in or plans to enroll in any concurrent drug, surgery and/or device study that may confound the results of this registry.

Registry Procedures

After the physician has determined that a patient meets all of the eligibility criteria, the physician will enroll the patient in the registry by completing the Patient Informed Consent or Data Release Consent Form process.

Once enrolled, patients will be followed at least for 24 months or until their discontinuation from the registry.

Follow-up visits will occur according to clinical practice, approximately every 6 months after the first visit post-implant.

Adverse events and/or device events will be reported as they occur.

Data collection will occur at the following time points:

* Enrollment Visit
* Baseline Visit
* Implant Visit
* Follow-up Visits (over a period of minimum two years)

The following follow-up visits are scheduled according to the clinical practice, approximately every 6 months for at least two years or till the closure of the registry.

Primary Objective The primary efficacy objective is to evaluate the change in seizure rate from baseline over 2 years following DBS implant.

Secondary Objectives

* To characterize the demographics of the population undergoing Medtronic® DBS™ Therapy for Epilepsy,
* To assess adverse events related to the device, implant procedure, and/or therapy.
* To characterize seizure type and severity.
* To characterize co-treatments.
* To assess the change in health-related quality of life following DBS by means of QOLIE-31 (Quality of life in epilepsy-31) and SF-36 (Short-form 36).
* To evaluate changes in depression score over time Exploratory objectives
* To assess use of health care resources specifically associated with epilepsy following DBS.
* To characterize DBS implant technique and device/feature utilization.
* To assess the factors that better predict the response level of the DBS therapy.

Sample Size Justification The purpose of the registry is essentially observational and exploratory; hence no sample size calculation was performed.

Safety objectives

* To assess adverse events
* To characterize the incidence of sudden unexpected death in epilepsy (SUDEP)

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the criteria of labeling indications of Medtronic® DBS™ Therapy for Epilepsy.
* Patient with diagnosis of refractory epilepsy as defined by 1981 ILAE (International League Against Epilepsy) classification, who have been implanted or will be implanted with Medtronic® DBS™ Therapy for Epilepsy.
* For both cohorts, completed at least two full consecutive months diary information on seizure type and frequency prior to DBS implant (seizure type should be classified at least as simple partial, complex partial, partial evolving to secondarily generalized seizures, and generalized). In regard to the prospective cohort, the patient will be conditionally enrolled at the enrolment visit, and the criterion will be reassessed at the baseline visit.
* Patient or patient's legally authorized representative able to understand and to provide written informed consent and/or authorization for access to and use of health information, as required by an institution's IRB/MEC or local law and regulations.

Exclusion Criteria:

* Incomplete and/or unreliable patient seizure diary based on the physician's judgment
* Patient is currently enrolled in or plans to enroll in any concurrent drug, surgery and/or device study that may confound the results of this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with refractory epilepsy characterized by partial-onset seizures, with or without secondary generalization
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2012-03-06 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Seizure rate | Participants will be followed for the duration of the registry, an expected average of 3 years
  Evaluate the change in seizure rate from baseline over 2 years following DBS implant.

SECONDARY OUTCOMES:
Seizure type and severity | Participants will be followed for the duration of the registry, an expected average of 3 years
  To characterize seizure type and severity
Depression score assessment | Participants will be followed for the duration of the registry, an expected average of 3 years
  To evaluate changes in depression score over time. BDI-II score is obtained by adding the score circled for each of the 21 items, the change of the BDI-II score is calculated as the difference between value at baseline phase and follow-up visits
Health Related Quality of Life (HRQoL) | Participants will be followed for the duration of the registry, an expected average of 3 years
  To assess the change in health-related quality of life following DBS by means of QOLIE-31 (Quality of life in epilepsy-31) and SF-36 (Short-form 36)
Adverse Events characterization | Participants will be followed for the duration of the registry, an expected average of 3 years
  To assess adverse events related to the device, implant procedure, and/or therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Boon, MD, Principal Investigator — Private
Locations (27):
- Medizinische Universität Wien, Vienna, Austria
- Belgium (2):
  - UZ Gent, Ghent
  - UZ K.U. Leuven, Leuven
- London Health Sciences Centre, London, Ontario, Canada
- University & Hospital of Tampere - Neurology and Rehabilitation, Tampere, Finland
- Germany (5):
  - Universitätsklinikum Bonn -AöR-, Bonn
  - University Hospital Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Klinikum der Universität München -Großhadern, Munich
  - University Hospital Tübingen, Tübingen
- Hungary (2):
  - Országos Idegtudományi Intézet / National Institute of Neurosciences, Budapest
  - University of Pécs Clinical Centre (PTE KK), Pécs
- Italy (3):
  - AZ. Ospedaliero-Universitario-Ospedali Riuniti, Ancona
  - AO Niguarda Ca' Granda, Milan
  - AO Santa Maria della Misericordia di Udine, Udine
- Netherlands (3):
  - SEIN Heemstede, Heemstede
  - Expertisecentrum Voor Epileptologie-Kempenhaeghe, Heeze
  - SEIN, Zwolle
- Poland (2):
  - Szpital Uniwersytecki w Krakowie - Neurology, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar de São João E.P.E., Porto
- Federal center of neurosurgery, Tyumen, Russia
- Sweden (3):
  - Karolinska University Hospital, Stockholm
  - Klinisk Neurovetenskap, Umeå
  - Uppsala Akademiska Hospital, Uppsala
- Frenchay Hospital, Bristol, United Kingdom

REFERENCES:
- [Derived] Peltola J, Colon AJ, Pimentel J, Coenen VA, Gil-Nagel A, Goncalves Ferreira A, Lehtimaki K, Ryvlin P, Taylor RS, Ackermans L, Ardesch J, Bentes C, Bosak M, Burneo JG, Chamadoira C, Elger CE, Eross L, Fabo D, Faulkner H, Gawlowicz J, Gharabaghi A, Iacoangeli M, Janszky J, Jarvenpaa S, Kaufmann E, Kho KH, Kumlien E, Laufs H, Lettieri C, Linhares P, Noachtar S, Parrent A, Pataraia E, Patel NK, Peralta AR, Racz A, Campos AR, Rego R, Ricciuti RA, Rona S, Rouhl RPW, Schulze-Bonhage A, Schuurman R, Sprengers M, Sufianov A, Temel Y, Theys T, Van Paesschen W, Van Roost D, Vaz R, Vonck K, Wagner L, Zwemmer J, Abouihia A, Brionne TC, Gielen F, Boon PAJM; MORE Study Group. Deep Brain Stimulation of the Anterior Nucleus of the Thalamus in Drug-Resistant Epilepsy in the MORE Multicenter Patient Registry. Neurology. 2023 May 2;100(18):e1852-e1865. doi: 10.1212/WNL.0000000000206887. Epub 2023 Mar 16. PMID 36927882